CLINICAL TRIAL: NCT03012230
Title: A Phase 1 Study of PD-1 Inhibition With Pembrolizumab Combined With JAK2 Inhibition in Triple Negative Breast Cancer
Brief Title: Pembrolizumab and Ruxolitinib Phosphate in Treating Patients With Metastatic Stage IV Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1534; NCI-2016-02057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-006282 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Malignant Neoplasm in the Bone; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, ruxolitinib phosphate) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and ruxolitinib phosphate PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase I trial studies the side effects and best dose of ruxolitinib phosphate when given together with pembrolizumab in treating patients with stage IV triple negative breast cancer that has spread to other places in the body. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ruxolitinib phosphate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and ruxolitinib phosphate together may work better in treating patients with stage IV triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of ruxolitinib phosphate (ruxolitinib) (JAK2 inhibition) in combination with fixed dosing of pembrolizumab (anti PD-1) in patients with advanced/metastatic triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To determine the safety profile of pembrolizumab in combination with ruxolitinib.

II. To estimate clinical tumor response in women with TNBC treated with pembrolizumab in combination with ruxolitinib as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. To assess tumor response with immune related (ir)RECIST and associations with PDJ amplification, PD-L1, PD-L2, JAK2 and phosphorylated (p)STAT3 expression.

II. To determine the effect of combination targeted blockade on T- and B- cell immunity to breast cancer tumor antigens.

OUTLINE: This is a dose-escalation study of ruxolitinib phosphate.

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and ruxolitinib phosphate orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up every 3 or 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Metastatic (stage IV) triple negative breast cancer that has progressed after at least one prior chemotherapy regimen in the metastatic setting or refusal of chemotherapy in the metastatic setting; non-measurable disease (i.e. bone metastases) is permitted
* Histological confirmation of triple negative breast cancer defined as:

  * Her2/neu by fluorescence in situ hybridization (FISH) (ratio =< 1.8) or immunohistochemistry (IHC) (0 or 1+)
  * Estrogen receptor (ER) and progesterone receptor (PR) expression < 10%
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 7 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 7 days prior to registration)
* Total bilirubin =< 1.5 x upper limit normal (ULN) (obtained =< 7 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN or < 5 x ULN if organ involvement (obtained =< 7 days prior to registration)
* Alkaline phosphatase < 5 x ULN (obtained =< 7 days prior to registration)
* Serum creatinine =< 2 x ULN or 24 hour creatinine (Cr) clearance > 60 ml/min (obtained =< 7 days prior to registration)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to provide informed written consent and be able to adhere to the study visit schedule and other protocol requirements
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes
* Has existing archived tissue and is willing to consent to providing sample for correlative research purposes
* Female subjects of childbearing potential should have a negative serum pregnancy =< 7 days prior to registration
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy; Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Radiographic or clinically measurable evidence of disease progression
* Prior therapy with atezolizumab is acceptable providing that all atezolizumab-related toxicities have resolved

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, known positive for active infectious hepatitis, type A, B or C (past infection allowed), or psychiatric illness/social situations that would limit compliance with study requirements; Note: ongoing infection controlled on antibiotics/antifungal/antiviral medications are allowed
* Any of the following prior therapies:

  * Cytotoxic chemotherapy =< 14 days prior to registration
  * Immunotherapy =< 14 days prior to registration
  * Biologic therapy (i.e. antibody therapies) =< 28 days prior to registration
  * Radiation therapy =< 14 days prior to registration
  * Targeted therapies (i.e. PARP inhibitors, =< 7 days or 5 half-lives whichever is shorter)
  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 14 days prior to registration
* Active uncontrolled central nervous system (CNS) metastases
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Hypersensitivity to ruxolitinib or any of its excipients
* Major surgery =< 28 days prior to registration; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Clinically significant heart disease, including the following:

  * Active severe angina pectoris prior to registration
  * Acute myocardial infarction prior to registration
  * New York Heart Association classification IV cardiovascular disease or symptomatic class III disease
  * Note: patients with any of the above may be allowed after discussion amongst the investigators including the principal investigator
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) =< 4 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline level) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy who has not recovered (i.e., =< grade 1 or at baseline level) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with pembrolizumab, nivolumab, avelumab, durvalumab
* Has received a live vaccine within 30 days of planned start of registration; Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Evidence of pericardial involvement with metastatic breast cancer (effusion, pericardial thickening)
* Radiographic evidence of pulmonary lymphangitic spread of metastatic breast cancer
* Evidence of bilateral pleural involvement with metastatic breast cancer (effusions, pleural thickening)
* Elevated serum lactate dehydrogenase level (LDH > laboratory ULN) associated with any clinical or radiographic evidence of intrathoracic metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 21 days
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients. Assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Incidence of adverse events | Up to 28 days after last dose of study drug
  Assessed by NCI CTCAE version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by cohort and overall). Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The rate of grade 3 or higher non-hematologic adverse events, and the rate of grade 4 or higher adverse event (hematologic and non-hematologic) will be computed each with a 95% exact binomial confidence.

SECONDARY OUTCOMES:
Best response | Up to 2 years
  Defined as best objective status recorded from the start of the treatment until disease progression/recurrence. Assessed by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by dose level).

OTHER OUTCOMES:
Assessment of PDJ amplification, PD-L1, PD-L2, JAK2 expression and pSTAT3 | Up to 2 years
  Will be explored for any associations with response to therapy. Statistical analysis of each biomarker will be primarily descriptive. Continuous biomarker levels will be explored in a graphical manner including mean plots and plots of change and percent change from baseline and other summary measures. Any potential relationships between the baseline level or change in the level of each biomarker and clinical outcome such as overall response will be further analyzed using Wilcoxon rank sum tests or logistic regression methods, as appropriate. Association between a dichotomized biomarker and overall response will be assessed using a chi-squared test. Comparisons with 1-sided p-values =< 0.10 are considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Northfelt, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States